CLINICAL TRIAL: NCT04300907
Title: An Open-Label Trial of PEMF Therapy [Provant Infinity Therapy System] for Home Use in Postoperative Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBI.2020.002
Record Dates: First submitted 2020-02-21; First posted 2020-03-09 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Provant Infinity Therapy (Experimental): Open-label treatment with Provant Infinity Therapy
  Interventions: Device: Provant Infinity Therapy System

INTERVENTIONS:
Device: Provant Infinity Therapy System — Treatment with the Provant Infinity Therapy System, PEMF device

SUMMARY:
A study of the use of the Provant Infinity Therapy System when treatment is administered 30 minutes twice daily for 8-weeks (56 days ± 3 days) at home for postoperative pain.

DETAILED DESCRIPTION:
This is an 8-week (56 days ± 3 days), multi-center, open label clinical trial conducted on subjects with chronic postoperative pain.

Eligible subjects will include those between 22 and 80 years of age with chronic postoperative pain at least 60 days following surgery.

At the Screening Visit, eligible subjects will have an average weekly pain score, over the last 7 days of ≥4 and <9 based on the 11-point NPRS (0-10) and will verbally confirm they have chronic postoperative pain from surgery ≥ 60 days prior . After signing Informed Consent and verifying subject eligibility for the trial (including a pain score assessment using the NPRS), subjects will have demographic information, medical/surgical history and medication use reviewed and recorded. An abbreviated physical examination, including height and weight, will be performed. A urine pregnancy test will be performed on women of childbearing potential.

Screening and Baseline (Day 0) / Enrollment may occur on the same day. During the Enrollment visit, subjects will receive study device training and be dispensed a study device with instructions to self-treat twice daily (morning and evening; 8am ± 2 hours and 8pm ± 2 hours) for 8 weeks (56 days ± 3 days).

If Screening and Enrollment are not on the same day, subjects returning to the clinic for Baseline (Day 0) will have an additional review of eligibility, medical history, adverse events and concomitant medications prior to device training and dispensation.

Subjects will receive a telephone call at Week 2 / Day 14 (±3 days). During the phone call subjects will have adverse events, and concomitant medications reviewed. Average weekly pain score (using the NPRS), Patient Global Impression (PGI), Treatment Satisfaction and Device Use questions will be captured.

Subjects will receive a telephone call at Week 4 / Day 28 (±3 days). During the phone, call subjects will have adverse events, and concomitant medications reviewed. Average weekly pain score (using the NPRS), Patient Global Impression (PGI), Treatment Satisfaction and Device Use questions will be captured.

Subjects will receive a telephone call at Week 6 / Day 42 (±3 days). During the phone, call subjects will have adverse events, and concomitant medications reviewed. Average weekly pain score (using the NPRS), Patient Global Impression (PGI), Treatment Satisfaction and Device Use questions will be captured.

At the Week 8 / Day 56 (±3 days) End of Study Visit, subjects will have adverse events and concomitant medications reviewed. Average weekly pain score (using the NPRS), Patient Global Impression (PGI), Treatment Satisfaction and Device Use and Feedback questions will be captured and the study device will be returned.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is ≥ 60 days postoperative. 2. Subject's average chronic postoperative pain over the preceding week is ≥4 and <9, based on the 11-point NPRS (0-10) at the Screening Visit.

  3. Subject's age is greater than or equal to 22 years and less than 80 years of age.

  4. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.

  5. Female subjects must be postmenopausal, surgically sterile, abstinent, or, if of childbearing potential, practicing (or agrees to practice) an effective method of birth control if they are sexually active for the duration of the study. Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization.

Exclusion Criteria:

* 1. Subject has a history of previous solid organ transplant or severe renal disease (i.e. estimated creatinine clearance <30 mL/min).

  2. Subject has previous or current history of primary or tertiary hyperparathyroidism, hypercalcemia, psychiatric disorder, alcohol dependency, Hepatitis B or C, or HIV infection.

  3. According to the judgment of the Investigator, subject has clinically significant cardiovascular disease within 6 months prior to screening (unstable or poorly controlled hypertension, transient ischemic attack, myocardial infarction, unstable angina, arrhythmia, cardiac surgery, stent placement or angioplasty, or congestive heart failure).

  4. Subject has a history of any uncontrolled medical illness that, in the investigator's judgment, places the subject at unacceptable risk for enrollment in a research trial with pulsed electromagnetic field therapy.

  5. Subject requires or anticipates the need for surgery (other than minor outpatient surgical procedures, such as dental or minor cosmetic procedures) or extended travel during the treatment period.

  6. Subject has received any investigational drug or device within 30 days prior to the Screening Visit.

  7. Subject has a history of malignancy within the past 5 years in the treatment area.

  8. Subject has severe mental health or psychiatric disorder that would interfere with study performance and/or assessments in the opinion of the Investigator.

  9. Subject has a known history of drug or alcohol abuse within one year prior to the Screening Visit.

  10. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).

  11. Subject is currently pregnant or planning to become pregnant prior to Week 8.

  12. Subject is unwilling or unable to follow study instructions or comply with the treatment regimen, diary documentation, and study visits.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Device Use Questionnaire | Week 8
  4 question questionnaire on device usage (total of all responses will be counted at the end of the study); response will require a "Yes" or "No" answer

SECONDARY OUTCOMES:
Device Feedback Questionnaire | Week 8
  5 question questionnaire about the study device; device use questions will be open text, "Yes" or "No" answers or rated from "Extremely Easy/Extremely Comfortable" to "Extremely Difficult/Extremely Uncomfortable"
Numeric Pain Rating Scale (NPRS) | Weeks 2, 4, 6 and 8
  11-point numerical rating scale for pain (0 = no pain to 10 = worst possible pain)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Physician's Research Group, Mesa, Arizona
  - Valley Clinical Research, Northridge, California
  - Lake Internal Medicine Associates, Eustis, Florida
  - Palm Research Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No